CLINICAL TRIAL: NCT03296306
Title: Four Cycles of Cisplatin-Based Chemotherapy in Metastatic Urothelial Carcinoma Compared to Six Cycles: Randomized Phase III Trial - FOCUS Study -
Brief Title: Four Cycles Versus Six Cycles of Cisplatin-based Chemotherapy in Metastatic Urothelial Carcinoma
Acronym: FOCUS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Jae-Lyun Lee, Associated Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCSG GU16-02
Record Dates: First submitted 2016-08-22; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Bladder Cancer; Ureter Cancer; Urethral Cancer; Transitional Cell Carcinoma
Keywords: urothelial carcinoma; cisplatin; first-line chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6 cycles arm (Active Comparator): Patients without evidence of disease progression or unacceptable toxicities after completion of two or four treatment cycles of cisplatin based chemotherapy (GP, GP-S, MVAC, HD-MVAC with GCSF) were randomly assigned to receive additional two to four cycles of chemotherapy (totally six cycles)
  Interventions: Drug: Treatment duration of cisplatin based chemotherapy
- 4 cycles arm (Experimental): Patients without evidence of disease progression or unacceptable toxicities after completion of two or four treatment cycles of cisplatin based chemotherapy (GP, GP-S, MVAC, HD-MVAC with GCSF) were randomly assigned to receive additional zero to two cycles of chemotherapy (totally four cycles)
  Interventions: Drug: Treatment duration of cisplatin based chemotherapy

INTERVENTIONS:
Drug: Treatment duration of cisplatin based chemotherapy — * GP regimen: Gemcitabine (1000 mg/m2 D1, D8), Cisplatin (60 mg/m2 D1), every 3 weeks
  * GP-S regimen: Gemcitabine (1000 mg/m2 D1, D8), Cisplatin (35 mg/m2 D1,D 2 or D8), every 3 weeks
  * MVAC regimen: Methotrexate (30 mg/m2 IV bolus, D1, 15, 22), Vinblastine (3 mg/m2 IV bolus, D2, 15, 22), Doxorubicin (30 mg/m2 IV bolus D2), Cisplatin (70 mg/m2 D2), every 4 weeks
  * HD-MVAC with GCSF regimen: Methotrexate (30 mg/m2 IV bolus, D1), Vinblastine (3 mg/m2 IV bolus, D2), Doxorubicin (30 mg/m2 IV bolus D2), Cisplatin (70 mg/m2 D2), G-CSF (240 ug/m2 SC, D4-10), every 2 weeks

SUMMARY:
The objective is to show non-inferiority of overall survival between four cycles and six cycles of first-line cisplatin based chemotherapy to determine the optimal duration of chemotherapy in patients with advanced urothelial carcinoma.

DETAILED DESCRIPTION:
Urothelial carcinoma is the fifth most common cancer in men and seventh among women all around the world. Although a complete surgical resection with or without perioperative treatment is the most effective way to offer a potentially curative therapy to patients with these cancers, 25% of the patients initially present with locally or systemically advanced disease. Systemic chemotherapy is the only current modality that provides the potential for a long-term survival in patients with advanced or metastatic urothelial disease.

Cisplatin based combination chemotherapies such as GP, GP-S, MVAC, and dose dense MVAC with G-CSF supports are regarded as a backbone treatment for patients with advanced bladder cancer on the basis of the results from previous studies.

However, there is no consensus on appropriate number of chemotherapy cycles. In phase III trial comparing MVAC with GP, patients were treated with 6 cycles (every 4 weeks) of chemotherapy. In another phase III trial comparing MVAC with HD-MVAC, there is no pre-determined number of cycles, but the median number of cycles were 4 for MVAC and 6 for HD-MVAC.

However, it is hard to complete six or more cycles of cisplatin based chemotherapy due to cumulative toxicities of cisplatin such as neuropathy and development of resistance. The median age of patients with urothelial cancer is 70 years old and significant proportion of the patients already showed impaired performance status (ECOG PS ≥2).

There has already been reported in several trials of NSCLC, which showed that 4 cycles of chemotherapy containing cisplatin has no significant differences in survival or QoL with lower incidences of toxicities compared with 6 cycles of chemotherapy.

The objective of this trial is to assess whether there is any difference in OS between patients who are treated with four cycles of cisplatin based chemotherapy and patients who are treated with 6 cycles of chemotherapy to determine the optimal duration of chemotherapy in patients with advanced urothelial cancer.

ELIGIBILITY:
Inclusion criteria:

1. Patients with histologically or cytologically confirmed urothelial cancer
2. Unresectable locally advanced (T3b, N2-3), metastatic (M1), or recurrent disease
3. Age 18 years or older
4. Eastern Cooperative Oncology Group performance status 0-1
5. Not progressed disease status after 2 or 4 cycles of platinum-based chemotherapy
6. Adequate organ and bone marrow function for chemotherapy
7. No history of radiation therapy, or radiation field within 25% of whole marrow would be allowed. If patients underwent radiation therapy in entire pelvis, they are excluded to this study. Patients should discontinue radiation therapy at least 4 weeks before enrollment, and the patients should be recovered from radiation therapy associated adverse events.
8. Women should use contraceptive medication for 6 months after the end of the study or she would be post-menopause status. Men should consent with the contraception for 6 months after the end of the study or he would be infertile.
9. Patients should sign a written informed consent before study entry.

Exclusion Criteria:

1. Histologic types other than urothelial cell carcinoma should be excluded. However, urothelial cell types combined with squamous or glandular features are allowed.
2. Patients who showed progressed disease status after 2 or 4 cycles of platinum-based chemotherapy, cannot be treated with additional chemotherapy due to adverse events, or already undertook with reduced dose of more than 50%
3. Presence or history of CNS metastasis
4. Prior systemic chemotherapy (But prior intravesical chemotherapy or immunotherapy was allowed, and recurrent disease after adjuvant or neoadjuvant cisplatin-based systemic chemotherapy is allowed if the last chemotherapy was administered 1 year or more before the patient enrollment)
5. Peripheral sensory neuropathy grade 2 or worse according to NCI CTCAE
6. History of treatment with drugs of another clinical trial within 30 days before enrollment.
7. Concomitant severe medical, surgical, or psychiatric disease or problems which can affect the results of the clinical trial or have possibilities of unexpected medical problems caused be the drug of clinical trial
8. History of another malignancy (but treated malignancy at least two years before enrollment were allowed, and cured non-melanoma skin cancer, any cured in-situ carcinoma, clinically insignificant localized prostate cancer, or papillary thyroid carcinoma are allowed even diagnosed less than 2 years before enrollment).
9. Pregnant or lactating women, women of childbearing potential not employing adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2016-09; Primary Completion 2021-08 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Overall survival is defined as the time from enrollment of study until death from any cause (or date of last follow-up for patients still alive)

SECONDARY OUTCOMES:
Progression free survival | Every 6-8 weeks, from date of enrollment until the date of first documented progression
  PFS is defined as the time from enrollment of study until either first documentation of RECIST-defined disease progression or death due to any cause, whichever come first.
Tumor response rate | Every 6-8 weeks, assess the tumor response from date of enrollment
  Tumor response rate is defined as the proportion of patients with a complete response (CR) or partial response (PR) among patients with evaluable lesions for response of RECIST.
safety using NCI Common Terminology Criteria for Adverse Events (version 4.03) | Every 2-4 weeks, from date of enrollment until 30th days of last cycles treatment or initation of new regimen
  Toxicity profiles will be evaluated every cycle with physical examination, vital signs, performance status, CBC, and serum chemistry using NCI Common Terminology Criteria for Adverse Events version 4.03.
Quality of life composite score of EORTC-QoL-C30 and EORTC CIPN20 | 0-1 week, 12-18 week, 24-34 week after enrollment
  Investigators measured Quality of life using EORTC-QoL-C30 and EORTC CIPN20 at the time of enrollment, 12-18 weeks, and 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Lyun Lee, MD., PhD., Principal Investigator — Asan Medical Center
Locations (19):
- South Korea (19):
  - Kwonoh Park, Yangsan, Gyeongsangnam-do
  - Hallym University Medical Center, Hallym University College of Medicine, Anyang
  - Fatima Hospital, Daegu
  - Keimyeong University Dongsan Medical Center, Daegu
  - Chungnam University Hospital, Daejeon
  - National Health Insurance Service Ilsan Hospital, Goyang
  - Gil Medical Center, Incheon
  - Inje University Haeundae Paik Hospital, Pusan
  - Kosin University Hospital, Pusan
  - Pusan National University Hospital, Pusan National University School of Medicine, Pusan
  - Asan Medical Center, Seoul
  - Chung Ang University Hospital, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Kangbuk Samsung Hospital, Sungkyunkwan University School of Medicine, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Cancer Research Institute, Seoul National University College of Medicine, Seoul
  - VHS medical center, Seoul
  - Yonsei Cancer Center, Seoul
  - St. Vincent's Hospital, The Catholic University of Korea, Suwon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cheng T. Systemic therapy for unresectable and metastatic transitional cell carcinoma of the urothelium: first-line and beyond. Curr Opin Support Palliat Care. 2008 Sep;2(3):153-60. doi: 10.1097/SPC.0b013e328309c72c. PMID 18685414
- [Result] von der Maase H, Hansen SW, Roberts JT, Dogliotti L, Oliver T, Moore MJ, Bodrogi I, Albers P, Knuth A, Lippert CM, Kerbrat P, Sanchez Rovira P, Wersall P, Cleall SP, Roychowdhury DF, Tomlin I, Visseren-Grul CM, Conte PF. Gemcitabine and cisplatin versus methotrexate, vinblastine, doxorubicin, and cisplatin in advanced or metastatic bladder cancer: results of a large, randomized, multinational, multicenter, phase III study. J Clin Oncol. 2000 Sep;18(17):3068-77. doi: 10.1200/JCO.2000.18.17.3068. PMID 11001674
- [Result] Sternberg CN, de Mulder P, Schornagel JH, Theodore C, Fossa SD, van Oosterom AT, Witjes JA, Spina M, van Groeningen CJ, Duclos B, Roberts JT, de Balincourt C, Collette L; EORTC Genito-Urinary Cancer Group. Seven year update of an EORTC phase III trial of high-dose intensity M-VAC chemotherapy and G-CSF versus classic M-VAC in advanced urothelial tract tumours. Eur J Cancer. 2006 Jan;42(1):50-4. doi: 10.1016/j.ejca.2005.08.032. Epub 2005 Dec 5. PMID 16330205
- [Result] Loehrer PJ Sr, Einhorn LH, Elson PJ, Crawford ED, Kuebler P, Tannock I, Raghavan D, Stuart-Harris R, Sarosdy MF, Lowe BA, et al. A randomized comparison of cisplatin alone or in combination with methotrexate, vinblastine, and doxorubicin in patients with metastatic urothelial carcinoma: a cooperative group study. J Clin Oncol. 1992 Jul;10(7):1066-73. doi: 10.1200/JCO.1992.10.7.1066. PMID 1607913
- [Result] Kim YR, Lee JL, You D, Jeong IG, Song C, Hong B, Hong JH, Ahn H. Gemcitabine plus split-dose cisplatin could be a promising alternative to gemcitabine plus carboplatin for cisplatin-unfit patients with advanced urothelial carcinoma. Cancer Chemother Pharmacol. 2015 Jul;76(1):141-53. doi: 10.1007/s00280-015-2774-z. Epub 2015 May 23. PMID 26001531
- [Result] Park JO, Kim SW, Ahn JS, Suh C, Lee JS, Jang JS, Cho EK, Yang SH, Choi JH, Heo DS, Park SY, Shin SW, Ahn MJ, Lee JS, Yun YH, Lee JW, Park K. Phase III trial of two versus four additional cycles in patients who are nonprogressive after two cycles of platinum-based chemotherapy in non small-cell lung cancer. J Clin Oncol. 2007 Nov 20;25(33):5233-9. doi: 10.1200/JCO.2007.10.8134. PMID 18024869